CLINICAL TRIAL: NCT02453711
Title: Investigation of Safety and Efficacy of Once-daily Semaglutide in Obese Subjects Without Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9536-4153; 2014-001540-38 (EudraCT Number); U1111-1155-4660 (Other: WHO)
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Results first posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity | interventions — semaglutide; Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (16):
- Sema 0.05 mg (Experimental): Dose 0.05 mg
  Interventions: Drug: semaglutide
- Sema 0.1 mg (Experimental): Dose 0.05 or 0.1 mg with dose escalation every fourth week
  Interventions: Drug: semaglutide
- Sema 0.2 mg (Experimental): Dose 0.05, 0.1 or 0.2 mg with dose escalation every fourth week
  Interventions: Drug: semaglutide
- Sema 0.3 mg (Experimental): Dose 0.05, 0.1, 0.2 or 0.3 mg with dose escalation every fourth week
  Interventions: Drug: semaglutide
- Sema 0.4 mg (Experimental): Dose 0.05, 0.1, 0.2, 0.3, or 0.4 mg with dose escalation every fourth week
  Interventions: Drug: semaglutide
- Sema 0.3 mg (fast dose escalation) (Experimental): Dose 0.05, 0.1, 0.2 or 0.3 mg with dose escalation every second week
  Interventions: Drug: semaglutide
- Sema 0.4 mg (fast dose escalation) (Experimental): Dose 0.05, 0.1, 0.2, 0.3, or 0.4 mg with dose escalation every second week
  Interventions: Drug: semaglutide
- Lira 3.0 mg (Active Comparator): Dose 0.6, 1.2, 1.8, 2.4, 3.0 mg with dose escalation every week
  Interventions: Drug: liraglutide
- Placebo Sema 0.05 mg (Placebo Comparator): Placebo arm matching active arm Sema 0.05 mg
  Interventions: Drug: placebo
- Placebo Sema 0.1 mg (Placebo Comparator): Placebo arm matching active arm Sema 0.1 mg
  Interventions: Drug: placebo
- Placebo Sema 0.2 mg (Placebo Comparator): Placebo arm matching active arm Sema 0.2 mg
  Interventions: Drug: placebo
- Placebo Sema 0.3 mg (Placebo Comparator): Placebo arm matching active arm Sema 0.3 mg
  Interventions: Drug: placebo
- Placebo Sema 0.4 mg (Placebo Comparator): Placebo arm matching active arm Sema 0.4 mg
  Interventions: Drug: placebo
- Placebo Sema 0.3 mg (fast dose escalation) (Placebo Comparator): Placebo arm matching active arm Sema 0.3 mg (fast dose escalation)
  Interventions: Drug: placebo
- Placebo Sema 0.4 mg (fast dose escalation) (Placebo Comparator): Placebo arm matching active arm Sema 0.4 mg (fast dose escalation)
  Interventions: Drug: placebo
- Placebo Lira 3.0 mg (Placebo Comparator): Placebo arm matching active arm Lira 3.0 mg
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: semaglutide — Once-daily subcutaneous (s.c., under the skin) administration with dose escalation.
  Arms: Sema 0.05 mg; Sema 0.1 mg; Sema 0.2 mg; Sema 0.3 mg; Sema 0.3 mg (fast dose escalation); Sema 0.4 mg; Sema 0.4 mg (fast dose escalation)
Drug: liraglutide — Once-daily subcutaneous (s.c., under the skin) administration with dose escalation.
  Arms: Lira 3.0 mg
Drug: placebo — Once-daily subcutaneous (s.c., under the skin) administration.
  Arms: Placebo Lira 3.0 mg; Placebo Sema 0.05 mg; Placebo Sema 0.1 mg; Placebo Sema 0.2 mg; Placebo Sema 0.3 mg; Placebo Sema 0.3 mg (fast dose escalation); Placebo Sema 0.4 mg; Placebo Sema 0.4 mg (fast dose escalation)

SUMMARY:
This trial is conducted globally. The aim of this trial is to investigate safety and efficacy of once-daily semaglutide in obese subjects without diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria: - Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial - Male or female, age 18 years or older at the time of signing inform consent - Body mass index (BMI) equal or above 30.0 kg/m^2 at the screening visit - At least one unsuccessful weight loss attempt per investigator judgement Exclusion Criteria: - A HbA1c (glycosylated haemoglobin) equal to or above 6.5% at screening or diagnosed with type 1 or type 2 diabetes mellitus - Treatment with glucose lowering agent(s) within 90 days before screening - Screening calcitonin equal to or above 50 ng/L (pg/mL) - Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2 - History of pancreatitis (acute or chronic) - Obesity induced by endocrine disorders (e.g. Cushing Syndrome) - Treatment with any medication within 90 days before screening that based on investigator's judgement may cause significant weight change - Previous surgical treatment for obesity (liposuction and/or abdominoplasty performed 1 year before screening is allowed) - History of major depressive disorder within 2 years before randomisation - Any lifetime history of a suicidal attempt - Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using an adequate contraceptive method (adequate contraceptive measures as required by local regulation or practice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 957 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (66):
- United States (21):
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Golden, Colorado
  - Novo Nordisk Investigational Site, Waterbury, Connecticut
  - Novo Nordisk Investigational Site, Washington D.C., District of Columbia
  - Novo Nordisk Investigational Site, Crystal River, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, Elkridge, Maryland
  - Novo Nordisk Investigational Site, Rochester, New York
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Wadsworth, Ohio
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Bristol, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Round Rock, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Arlington, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
- Australia (5):
  - Novo Nordisk Investigational Site, Camperdown, New South Wales
  - Novo Nordisk Investigational Site, Merewether, New South Wales
  - Novo Nordisk Investigational Site, St Leonards, New South Wales
  - Novo Nordisk Investigational Site, Heidelberg Heights, Victoria
  - Novo Nordisk Investigational Site, Melbourne, Victoria
- Belgium (5):
  - Novo Nordisk Investigational Site, Brussels
  - Novo Nordisk Investigational Site, Edegem
  - Novo Nordisk Investigational Site, Leuven
  - Novo Nordisk Investigational Site, Liège
  - Novo Nordisk Investigational Site, Mons
- Canada (8):
  - Novo Nordisk Investigational Site, Calgary, Alberta
  - Novo Nordisk Investigational Site, Surrey, British Columbia
  - Novo Nordisk Investigational Site, Moncton, New Brunswick
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, Hamilton, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Montreal, Quebec
  - Novo Nordisk Investigational Site, Québec
- Germany (6):
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Duisburg
  - Novo Nordisk Investigational Site, Leipzig
  - Novo Nordisk Investigational Site, Saint Ingbert-Oberwürzbach
  - Novo Nordisk Investigational Site, Stuttgart
  - Novo Nordisk Investigational Site, Wangen
- Israel (6):
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Kfar Saba
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Tel Aviv
  - Novo Nordisk Investigational Site, Tel Litwinsky
- Russia (7):
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Penza
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Tyumen
  - Novo Nordisk Investigational Site, Voronezh
  - Novo Nordisk Investigational Site, Yaroslavl
- United Kingdom (8):
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Cambridge
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, Liverpool
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Luton
  - Novo Nordisk Investigational Site, Norwich
  - Novo Nordisk Investigational Site, Rotherham

REFERENCES:
- [Background] Kolotkin RL, Williams VSL, Ervin CM, Williams N, Meincke HH, Qin S, von Huth Smith L, Fehnel SE. Validation of a new measure of quality of life in obesity trials: Impact of Weight on Quality of Life-Lite Clinical Trials Version. Clin Obes. 2019 Jun;9(3):e12310. doi: 10.1111/cob.12310. Epub 2019 Apr 16. PMID 30993900
- [Result] O'Neil PM, Birkenfeld AL, McGowan B, Mosenzon O, Pedersen SD, Wharton S, Carson CG, Jepsen CH, Kabisch M, Wilding JPH. Efficacy and safety of semaglutide compared with liraglutide and placebo for weight loss in patients with obesity: a randomised, double-blind, placebo and active controlled, dose-ranging, phase 2 trial. Lancet. 2018 Aug 25;392(10148):637-649. doi: 10.1016/S0140-6736(18)31773-2. Epub 2018 Aug 16. PMID 30122305
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 71 sites in 8 countries as follows: Australia: 5, Belgium: 5, Canada: 9, Germany: 6, Israel: 7, Russian Federation: 10, United Kingdom (UK):8, United States (US): 21. Along with this, recruitment of participants was planned at 3 sites (1 each in Germany, Russian Federation, and US), but where no participants were screened
Pre-assignment Details: Design:Participants were randomised to 1 of the 16 parallel treatment arms in a 6:1 ratio (active:placebo) to receive either:A)Semaglutide 0.05/0.1/0.2/0.3/0.4 mg; dose escalation every 4th week B)Semaglutide 0.3/0.4 mg; dose escalation every second week C)Liraglutide 3.0 mg;dose escalation every week D)Placebo;matching each of the active treatment
Groups:
- Semaglutide 0.05 mg: Participants received once daily semaglutide 0.05 mg subcutaneous (s.c.; under the skin) injections for 52 weeks.
- Semaglutide 0.1 mg: Participants received once daily semaglutide s.c. injections for 52 weeks. Dose escalation was done at every fourth week as following: 0.05 mg (week 1 to week 4) and 0.1 mg (week 5 to week 52).
- Semaglutide 0.2 mg: Participants received once daily semaglutide s.c. injections for 52 weeks. Dose escalation was done at every fourth week as following: 0.05 mg (week 1 to week 4), 0.1 mg (week 5 to week 8), and 0.2 mg (week 9 to week 52).
- Semaglutide 0.3 mg: Participants received once daily semaglutide s.c. injections for 52 weeks. Dose escalation was done at every fourth week as following: 0.05 mg (week 1 to week 4), 0.1 mg (week 5 to week 8), 0.2 mg (week 9 to week 12), and 0.3 mg (week 13 to week 52).
- Semaglutide 0.4 mg: Participants received once daily semaglutide s.c. injections for 52 weeks. Dose escalation was done at every fourth week as following: 0.05 mg (week 1 to week 4), 0.1 mg (week 5 to week 8), 0.2 mg (week 9 to week 12), 0.3 mg (week 13 to week 16), and 0.4 mg (week 17 to week 52).
- Semaglutide 0.3 mg (Fast Escalation): Participants received once daily semaglutide s.c. injections for 52 weeks. Dose escalation was done at every second week (fast escalation) as following: 0.05 mg (in weeks 1 and 2), 0.1 mg (in weeks 3 and 4), 0.2 mg (in weeks 5 and 6), and 0.3 mg (week 7 to week 52).
- Semaglutide 0.4 mg (Fast Escalation): Participants received once daily semaglutide s.c. injections for 52 weeks. Dose escalation was done at every second week (fast escalation) as following: 0.05 mg (in weeks 1 and 2), 0.1 mg (in weeks 3 and 4), 0.2 mg (in weeks 5 and 6), 0.3 mg (in weeks 7 and 8), and 0.4 mg (week 9 to week 52).
- Liraglutide 3.0 mg: Participants received once daily liraglutide s.c. injections for 52 weeks. Dose escalation was done at every week as following: 0.6 mg in week 1, 1.2 mg in week 2, 1.8 mg in week 3, 2.4 mg in week 4, and 3.0 mg from week 5 to week 52.
- Placebo Pool: Participants received once daily placebo s.c injections (matching each of the active treatment arms: semaglutide 0.05 mg, 0.1 mg, 0.2 mg, 0.3 mg or 0.4 mg (dose escalation every fourth week); semaglutide 0.3 mg or 0.4 mg (dose escalation every second week); liraglutide 3.0 mg (dose escalation every week)).
Period: Overall Study
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Started | 103 | 102 | 103 | 103 | 102 | 102 | 103 | 103 | 136
Full Analysis Set | 103 | 102 | 103 | 103 | 102 | 102 | 103 | 103 | 136
Safety Analysis Set | 103 | 102 | 103 | 103 | 102 | 102 | 103 | 103 | 136
Completed | 92 | 95 | 94 | 96 | 100 | 96 | 100 | 96 | 123
Not Completed | 11 | 7 | 9 | 7 | 2 | 6 | 3 | 7 | 13
Not completed — Withdrawal by Subject | 5 | 4 | 6 | 4 | 1 | 1 | 0 | 1 | 7
Not completed — Lost to Follow-up | 5 | 3 | 2 | 3 | 1 | 5 | 2 | 6 | 6
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Unclassified | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Overall number of baseline participants = full analysis set (FAS) which included all randomised participants. Number Analyzed = number of participants with available data.
Groups:
- Semaglutide 0.05 mg: Participants received once daily semaglutide 0.05 mg s.c. injections for 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool | Total
Number analyzed (Participants) | 103 | 102 | 103 | 103 | 102 | 102 | 103 | 103 | 136 | 957
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.97 (12.80) | 45.24 (12.62) | 44.37 (11.24) | 46.73 (12.02) | 48.37 (13.44) | 47.10 (12.05) | 46.07 (13.51) | 48.50 (11.22) | 46.42 (12.80) | 46.63 (12.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 66 | 66 | 66 | 66 | 66 | 67 | 67 | 88 | 619
  Male | 36 | 36 | 37 | 37 | 36 | 36 | 36 | 36 | 48 | 338
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 88 | 76 | 72 | 74 | 71 | 76 | 68 | 78 | 97 | 700
  Black or African American | 5 | 7 | 10 | 3 | 10 | 0 | 7 | 9 | 10 | 61
  Asian | 2 | 0 | 1 | 0 | 0 | 3 | 1 | 1 | 1 | 9
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
  Other | 0 | 1 | 0 | 3 | 1 | 1 | 0 | 1 | 2 | 9
  Not applicable | 8 | 17 | 20 | 22 | 19 | 22 | 25 | 14 | 24 | 171
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 6 | 13 | 4 | 6 | 3 | 6 | 7 | 55
  Not Hispanic or Latino | 96 | 86 | 93 | 79 | 90 | 82 | 91 | 93 | 117 | 827
  Not applicable | 4 | 9 | 4 | 11 | 8 | 14 | 9 | 4 | 12 | 75
Body weight [Mean (Standard Deviation); unit: Kilogram (Kg)] | 111.29 (23.17) | 111.31 (21.47) | 114.49 (24.53) | 111.51 (22.96) | 113.20 (26.42) | 108.11 (22.08) | 109.56 (21.33) | 108.71 (21.94) | 114.19 (25.37) | 111.48 (23.39)
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage (%) of HbA1c] — Population: Number Analyzed = number of participants in the FAS with available data. FAS included all randomised participants.
  Percentage (%) of HbA1c
    number analyzed (Participants) | 103 | 101 | 103 | 103 | 102 | 102 | 103 | 103 | 136 | 956
    (all) | 5.51 (0.35) | 5.45 (0.43) | 5.41 (0.39) | 5.51 (0.38) | 5.47 (0.42) | 5.48 (0.41) | 5.49 (0.42) | 5.53 (0.38) | 5.54 (0.38) | 5.49 (0.40)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: Millimoles per litre (mmol/L)] — Population: Number Analyzed = number of participants in the FAS with available data. FAS included all randomised participants.
  Millimoles per litre (mmol/L)
    number analyzed (Participants) | 103 | 102 | 103 | 103 | 101 | 102 | 103 | 103 | 136 | 956
    (all) | 5.48 (0.64) | 5.48 (0.55) | 5.41 (0.77) | 5.48 (0.73) | 5.40 (0.67) | 5.43 (0.64) | 5.54 (0.87) | 5.55 (0.73) | 5.50 (0.62) | 5.48 (0.69)

OUTCOME MEASURES:

1. Primary Outcome: Relative Change in Body Weight (%)
Description: Relative change from baseline (week 0) in body weight was evaluated at week 52. Analysis of in-trial data with missing observations imputed from the pooled placebo arms based on a jump to reference multiple (x1000) imputation (J2R-MI) approach. Week 52 responses were analysed using an analysis of covariance model with treatment, region and sex as factors and baseline body weight as covariate. In-trial observation period was defined as the period from randomisation to last contact with trial site.
Time Frame: Week 0, Week 52
Population: Overall number of participants analyzed = number of participants in the FAS who contributed to the analysis. FAS included all randomised participants.
Measure: Least Squares Mean (Standard Error); unit: Percentage (%) of body weight
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 92 | 96 | 94 | 95 | 100 | 95 | 100 | 96 | 123
Percentage (%) of body weight | -5.99 (0.85) | -8.62 (0.84) | -11.60 (0.85) | -11.17 (0.85) | -13.84 (0.83) | -11.38 (0.85) | -16.29 (0.83) | -7.76 (0.85) | -2.29 (0.74)
Statistical Analysis 1: Comparison: Semaglutide 0.05 mg vs Placebo Pool; J2R-MI: Analysis of in-trial data with missing observations imputed from the pooled placebo arms based on a jump to reference multiple (x1000) imputation (J2R-MI) approach. Week 52 responses were analysed using an analysis of covariance model with treatment, region and sex as factors and baseline body weight as covariate. Dunnett's method was used to adjust for multiple comparisons; Test type: Other; p = 0.0055, ANCOVA; Treatment difference (%-points) = -3.70, 95% CI 2-sided [-6.55 to -0.85], Standard Error of Mean 1.13 — Semaglutide 0.05 mg - placebo pool
Statistical Analysis 2: Comparison: Semaglutide 0.1 mg vs Placebo Pool; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, ANCOVA; Treatment difference (%-points) = -6.32, 95% CI 2-sided [-9.16 to -3.49], Standard Error of Mean 1.12 — Semaglutide 0.1 mg - placebo pool
Statistical Analysis 3: Comparison: Semaglutide 0.2 mg vs Placebo Pool; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, ANCOVA; Treatment difference (%-points) = -9.31, 95% CI 2-sided [-12.15 to -6.46], Standard Error of Mean 1.12 — Semaglutide 0.2 mg - placebo pool
Statistical Analysis 4: Comparison: Semaglutide 0.3 mg vs Placebo Pool; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, ANCOVA; Treatment difference (%-points) = -8.88, 95% CI 2-sided [-11.72 to -6.03], Standard Error of Mean 1.12 — Semaglutide 0.3 mg - placebo pool
Statistical Analysis 5: Comparison: Semaglutide 0.4 mg vs Placebo Pool; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, ANCOVA; Treatment difference (%-points) = -11.55, 95% CI 2-sided [-14.38 to -8.72], Standard Error of Mean 1.12 — Semaglutide 0.4 mg - placebo pool

2. Secondary Outcome: Participants With Weight Loss of ≥5% of Baseline Body Weight
Description: Presented results are percentage of participants who lost more than or equal to 5% of their baseline (week 0) body weight at week 52. Analysis of observed in-trial data with missing observations imputed from the pooled placebo arms based on a jump to reference multiple (x1000) imputation (J2R-MI) approach. Week 52 responses were analysed using a binary logistic regression model with treatment, region and sex as factors and baseline body weight as covariate. In-trial observation period was defined as the period from randomisation to last contact with trial site.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage (%) of participants
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 92 | 96 | 94 | 95 | 100 | 95 | 100 | 96 | 123
Percentage (%) of participants | 53.50 | 67.49 | 74.91 | 80.52 | 82.52 | 72.19 | 89.58 | 66.12 | 22.87

3. Secondary Outcome: Participants With Weight Loss of ≥10% of Baseline Body Weight
Description: Presented results are percentage of participants who lost more than or equal to 10% of their baseline (week 0) body weight at week 52. Analysis of observed in-trial data with missing observations imputed from the pooled placebo arms based on a jump to reference multiple (x1000) imputation (J2R-MI) approach. Week 52 responses were analysed using a binary logistic regression model with treatment, region and sex as factors and baseline body weight as covariate. In-trial observation period was defined as the period from randomisation to last contact with trial site.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage (%) of participants
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 92 | 96 | 94 | 95 | 100 | 95 | 100 | 96 | 123
Percentage (%) of participants | 18.94 | 36.57 | 55.95 | 57.76 | 64.61 | 58.45 | 71.91 | 33.98 | 10.08

4. Secondary Outcome: Change in Body Weight (kg)
Description: Change from baseline (week 0) in body weight was evaluated at week 52. Analysis of in-trial data with missing observations imputed from the pooled placebo arms based on a jump to reference multiple (x1000) imputation (J2R-MI) approach. Week 52 responses were analysed using an analysis of covariance model with treatment, region and sex as factors and baseline body weight as covariate. Results are based on the in-trial observation period which was defined as the period from randomisation to last contact with trial site.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Kilogram (kg)
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 92 | 96 | 94 | 95 | 100 | 95 | 100 | 96 | 123
Kilogram (kg) | -6.66 (0.94) | -9.34 (0.93) | -12.30 (0.93) | -12.45 (0.93) | -15.15 (0.92) | -12.54 (0.93) | -17.36 (0.92) | -8.47 (0.93) | -2.48 (0.82)

5. Secondary Outcome: Change in Waist Circumference
Description: Change from baseline (week 0) in waist circumference was evaluated at week 52. Analysis of in-trial data with missing observations imputed from the pooled placebo arms based on a jump to reference multiple (x1000) imputation (J2R-MI) approach. Week 52 responses were analysed using an analysis of covariance model with treatment, region and sex as factors and baseline waist circumference as covariate. Results are based on the in-trial observation period which was defined as the period from randomisation to last contact with trial site.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Centimetre (cm)
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 77 | 88 | 87 | 88 | 82 | 73 | 91 | 86 | 103
Centimetre (cm) | -6.11 (0.93) | -8.75 (0.90) | -11.02 (0.89) | -10.91 (0.89) | -12.31 (0.91) | -11.06 (0.95) | -14.88 (0.88) | -8.35 (0.89) | -3.47 (0.81)

6. Secondary Outcome: Change in Waist to Hip Circumference Ratio
Description: Change from baseline (week 0) in waist to hip circumference ratio was evaluated at week 52. Analysis of in-trial data with missing observations imputed from the pooled placebo arms based on a jump to reference multiple (x1000) imputation (J2R-MI) approach. Week 52 responses were analysed using an analysis of covariance model with treatment, region and sex as factors and baseline waist to hip circumference ratio as covariate. Results are based on the in-trial observation period which was defined as the period from randomisation to last contact with trial site.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Waist to hip circumference ratio
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 77 | 88 | 87 | 88 | 82 | 73 | 91 | 86 | 103
Waist to hip circumference ratio | -0.01 (0.01) | -0.02 (0.01) | -0.02 (0.01) | -0.03 (0.01) | -0.02 (0.01) | -0.02 (0.01) | -0.03 (0.01) | -0.02 (0.01) | -0.01 (0.00)

7. Secondary Outcome: Change in BMI
Description: Change from baseline (week 0) in body mass index (BMI) was evaluated at week 52. Analysis of in-trial data with missing observations imputed from the pooled placebo arms based on a jump to reference multiple (x1000) imputation (J2R-MI) approach. Week 52 responses were analysed using an analysis of covariance model with treatment, region and sex as factors and baseline BMI as covariate. Results are based on the in-trial observation period which was defined as the period from randomisation to last contact with trial site.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Kilogram per square meter (kg/m^2)
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 92 | 96 | 94 | 95 | 100 | 95 | 100 | 96 | 123
Kilogram per square meter (kg/m^2) | -2.37 (0.33) | -3.36 (0.33) | -4.38 (0.33) | -4.40 (0.33) | -5.40 (0.33) | -4.48 (0.33) | -6.21 (0.33) | -3.03 (0.33) | -0.88 (0.29)

8. Secondary Outcome: Change in HbA1c
Description: Change from baseline (week 0) in glycosylated haemoglobin (HbA1c) was evaluated at week 52. Analysis of in-trial data with missing observations imputed from the pooled placebo arms based on a jump to reference multiple (x1000) imputation (J2R-MI) approach. Week 52 responses were analysed using an analysis of covariance model with treatment, region and sex as factors and baseline HbA1c as covariate. Results are based on the in-trial observation period which was defined as the period from randomisation to last contact with trial site.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 77 | 88 | 87 | 87 | 82 | 75 | 91 | 85 | 103
Percentage of HbA1c | -0.13 (0.03) | -0.21 (0.03) | -0.28 (0.03) | -0.23 (0.03) | -0.29 (0.03) | -0.25 (0.03) | -0.34 (0.03) | -0.21 (0.03) | -0.01 (0.03)

9. Secondary Outcome: Change in FPG
Description: Change from baseline (week 0) in fasting plasma glucose (FPG) was evaluated at week 52. Analysis of in-trial data with missing observations imputed from the pooled placebo arms based on a jump to reference multiple (x1000) imputation (J2R-MI) approach. Week 52 responses were analysed using an analysis of covariance model with treatment, region and sex as factors and baseline FPG as covariate. Results are based on the in-trial observation period which was defined as the period from randomisation to last contact with trial site.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Millimoles per litre (mmol/L)
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 77 | 88 | 86 | 88 | 81 | 75 | 91 | 86 | 103
Millimoles per litre (mmol/L) | -0.29 (0.06) | -0.35 (0.06) | -0.40 (0.06) | -0.39 (0.06) | -0.43 (0.06) | -0.38 (0.06) | -0.51 (0.06) | -0.35 (0.06) | 0.01 (0.05)

10. Secondary Outcome: Change in Glycaemic Category (Normoglycaemia, Pre-diabetes, T2D)
Description: The categorisation of glycaemic status as described in the protocol was not aligned with the usual diagnosis criteria which require repeated testing of blood glucose to confirm the diagnosis and allows for the diagnosis to be made based on random glucose assessments and/or 2-hour glucose assessments during an oral glucose tolerance test. Therefore, data were not collected for this outcome measure.
Time Frame: Week 0, Week 52
Population: Data were not collected for this outcome measure.
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Change in SBP
Description: Change from baseline (week 0) in systolic blood pressure (SBP) was evaluated at week 52. Analysis of in-trial data with missing observations imputed from the pooled placebo arms based on a jump to reference multiple (x1000) imputation (J2R-MI) approach. Week 52 responses were analysed using an analysis of covariance model with treatment, region and sex as factors and baseline SBP as covariate. Results are based on the in-trial observation period which was defined as the period from randomisation to last contact with trial site.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Millimeters of mercury (mmHg)
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 91 | 96 | 94 | 95 | 100 | 95 | 100 | 96 | 123
Millimeters of mercury (mmHg) | -4.46 (1.20) | -5.76 (1.18) | -6.26 (1.19) | -6.41 (1.19) | -5.81 (1.16) | -6.07 (1.19) | -10.26 (1.16) | -5.45 (1.18) | -1.58 (1.04)

12. Secondary Outcome: Change in DBP
Description: Change from baseline (week 0) in diastolic blood pressure (DBP) was evaluated at week 52. Analysis of in-trial data with missing observations imputed from the pooled placebo arms based on a jump to reference multiple (x1000) imputation (J2R-MI) approach. Week 52 responses were analysed using an analysis of covariance model with treatment, region and sex as factors and baseline DBP as covariate. Results are based on the in-trial observation period which was defined as the period from randomisation to last contact with trial site.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Millimeters of mercury (mmHg)
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 91 | 96 | 94 | 95 | 100 | 95 | 100 | 96 | 123
Millimeters of mercury (mmHg) | -2.55 (0.84) | -2.65 (0.82) | -4.09 (0.83) | -2.98 (0.83) | -3.61 (0.80) | -2.20 (0.83) | -5.52 (0.80) | -2.70 (0.82) | -1.50 (0.73)

13. Secondary Outcome: Change in Lipids (Total Cholesterol, LDL Cholesterol, HDL Cholesterol, VLDL Cholesterol, Triglycerides and FFA)
Description: Change from baseline (week 0) in lipids (total cholesterol, low density lipoprotein (LDL) cholesterol, high density lipoprotein (HDL) cholesterol, very low density lipoprotein (VLDL) cholesterol and triglycerides) was evaluated at week 52. Analysis of in-trial data with missing observations imputed from the pooled placebo arms based on a jump to reference multiple (x1000) imputation (J2R-MI) approach. Week 52 responses were analysed using an analysis of covariance model with treatment, region and sex as factors and respective baseline lipid value as covariate. Results are based on the in-trial observation period which was defined as the period from randomisation to last contact with trial site. Free fatty acid (FFA) results are not presented as the values were considered invalid. The shipment of the samples to be tested for FFA was not as per the requirement.
Time Frame: Week 0, Week 52
Population: Overall number of participants analyzed = FAS which included all randomised participants. Number Analyzed = number of participants in the FAS who contributed to the analysis.
Measure: Least Squares Mean (Standard Error); unit: Millimoles per litre (mmol/L)
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 103 | 102 | 103 | 103 | 102 | 102 | 103 | 103 | 136
Millimoles per litre (mmol/L)
  Total cholesterol: number analyzed (Participants) | 77 | 88 | 87 | 87 | 82 | 74 | 91 | 85 | 102
  Total cholesterol | 0.96 (0.02) | 0.95 (0.01) | 0.93 (0.01) | 0.93 (0.01) | 0.93 (0.01) | 0.93 (0.02) | 0.92 (0.01) | 0.96 (0.01) | 0.97 (0.01)
  LDL cholesterol: number analyzed (Participants) | 72 | 87 | 86 | 85 | 82 | 72 | 89 | 82 | 100
  LDL cholesterol | 0.97 (0.02) | 0.93 (0.02) | 0.93 (0.02) | 0.92 (0.02) | 0.93 (0.02) | 0.92 (0.02) | 0.91 (0.02) | 0.95 (0.02) | 0.97 (0.02)
  HDL cholesterol: number analyzed (Participants) | 77 | 88 | 87 | 87 | 82 | 74 | 91 | 85 | 102
  HDL cholesterol | 0.99 (0.01) | 1.02 (0.01) | 1.02 (0.01) | 1.02 (0.01) | 1.00 (0.01) | 1.00 (0.02) | 1.01 (0.01) | 1.00 (0.01) | 1.00 (0.01)
  VLDL cholesterol: number analyzed (Participants) | 76 | 88 | 87 | 87 | 82 | 72 | 91 | 84 | 102
  VLDL cholesterol | 0.90 (0.03) | 0.89 (0.03) | 0.81 (0.03) | 0.85 (0.03) | 0.81 (0.03) | 0.87 (0.04) | 0.81 (0.03) | 0.91 (0.03) | 0.95 (0.03)
  Triglycerides: number analyzed (Participants) | 76 | 88 | 87 | 87 | 82 | 72 | 91 | 84 | 102
  Triglycerides | 0.89 (0.04) | 0.88 (0.03) | 0.81 (0.03) | 0.85 (0.03) | 0.80 (0.03) | 0.87 (0.04) | 0.80 (0.03) | 0.90 (0.03) | 0.95 (0.03)

14. Secondary Outcome: Change in hsCRP
Description: Change from baseline (week 0) in high-sensitivity C-reactive protein (hsCRP) was evaluated at week 52. Analysis of in-trial data with missing observations imputed from the pooled placebo arms based on a jump to reference multiple (x1000) imputation (J2R-MI) approach. Week 52 responses were analysed using an analysis of covariance model with treatment, region and sex as factors and baseline hsCRP as covariate. Results are based on the in-trial observation period which was defined as the period from randomisation to last contact with trial site.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Milligrams per decilitre (mg/dL)
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 77 | 88 | 87 | 87 | 82 | 74 | 91 | 85 | 102
Milligrams per decilitre (mg/dL) | 0.71 (0.07) | 0.65 (0.06) | 0.57 (0.05) | 0.66 (0.06) | 0.54 (0.05) | 0.58 (0.05) | 0.44 (0.04) | 0.72 (0.06) | 0.82 (0.07)

15. Secondary Outcome: Change in IWQoL Lite
Description: The planned analyses of the Impact of Weight on Quality of Life Lite (IWQoL-Lite) for Clinical Trials scores were not performed. The measure was still under development, and Novo Nordisk had not obtained a validated scoring of the instrument by the time of analysis of the trial results. Therefore, the total and subdomain scores on the IWQoL-Lite could not be provided.
Time Frame: Week 0, Week 52
Population: This outcome measure was not analysed.
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Change in SF-36
Description: Short Form-36 (SF-36) is a 36-item patient-reported survey of patient health that measures the participant's overall health-related quality of life (HRQoL). SF-36v2™ (acute version) questionnaire measured eight domains of functional health and well-being as well as two component summary scores (physical component summary (PCS) and mental component summary (MCS)). The 0-100 scale scores (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. In the metric of norm-based scores, 50 and 10 corresponds to the mean and standard deviation respectively of the 2009 U.S. general population. Change from baseline (week 0) in the domain scores and component summary (PCS and MCS) scores were evaluated at week 52. A positive change score indicates an improvement since baseline. Results are based on the in-trial observation period.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 27 | 23 | 20 | 31 | 33 | 22 | 24 | 31 | 37
Score on a scale
  Bodily pain | 1.85 (10.99) | 3.01 (6.41) | 4.27 (7.14) | 3.82 (7.11) | 5.16 (8.02) | 1.88 (9.25) | 5.11 (10.62) | 2.48 (7.46) | 1.21 (9.39)
  General health | 2.03 (5.98) | 2.51 (7.23) | 4.17 (6.52) | 1.20 (5.88) | 5.85 (7.62) | 5.85 (7.11) | 4.81 (10.33) | 3.95 (6.61) | 1.39 (8.98)
  Mental health | 0.42 (7.76) | 0.24 (6.57) | 2.82 (8.67) | -0.55 (6.48) | 2.47 (7.03) | 1.02 (6.93) | 1.64 (6.84) | 1.91 (6.06) | -0.38 (8.98)
  Physical functioning | 6.00 (6.92) | 4.67 (8.17) | 6.52 (5.91) | 4.75 (4.07) | 8.74 (7.66) | 7.27 (6.32) | 7.28 (6.27) | 6.79 (6.40) | 2.28 (7.56)
  Role-emotional | 3.31 (6.35) | -1.69 (6.61) | 1.17 (7.03) | 1.25 (7.47) | 2.24 (8.91) | 0.18 (3.69) | 2.11 (6.17) | 0.25 (5.01) | 0.63 (5.30)
  Role-physical | 3.45 (8.24) | 4.37 (10.23) | 7.35 (8.85) | 3.40 (5.43) | 4.53 (7.45) | 7.12 (8.21) | 5.51 (8.49) | 5.37 (6.82) | 1.52 (9.47)
  Social functioning | 0.81 (6.54) | 0.71 (7.04) | 1.36 (7.69) | -0.88 (8.81) | 2.81 (9.65) | 2.23 (7.07) | -0.91 (11.10) | 0.35 (5.62) | -0.29 (7.71)
  Vitality | 1.73 (7.61) | 5.16 (11.08) | 8.90 (8.61) | 3.22 (6.42) | 9.37 (9.75) | 5.96 (7.94) | 7.02 (9.35) | 4.83 (10.84) | 3.38 (10.21)
  Physical component summary | 4.16 (7.70) | 5.51 (8.04) | 7.14 (6.38) | 4.70 (4.67) | 7.67 (6.93) | 7.54 (8.29) | 7.28 (8.54) | 6.21 (5.68) | 2.29 (9.33)
  Mental component summary | 0.25 (5.94) | -1.15 (6.67) | 1.45 (8.54) | -1.10 (7.79) | 1.97 (8.26) | -0.25 (6.66) | 0.20 (7.13) | -0.26 (5.69) | -0.05 (6.67)

17. Secondary Outcome: Participants With Change in Concomitant Medications (Antihypertensive and Lipid-lowering Medications)
Description: Participants' status on receiving concomitant medication (antihypertensive and lipid-lowering medications) at week 0 (yes/no) and week 52 (decreased, no change, increased or missing) are presented. Results are based on the on-treatment observation period which was defined as the period from first trial product administration to last trial product administration.
Time Frame: Week 0, Week 52
Population: Overall number of participants analyzed = FAS which included all randomised participants. Number Analyzed = number of participants in the FAS with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 103 | 102 | 103 | 103 | 102 | 102 | 103 | 103 | 136
Participants
  Week 0: Antihypertensive medication (Yes) | 37 | 31 | 28 | 31 | 36 | 32 | 29 | 36 | 50
  Week 0: Antihypertensive medication (No) | 66 | 71 | 75 | 72 | 66 | 70 | 74 | 67 | 86
  Week 52: Antihypertensive medication (Decreased): number analyzed (Participants) | 77 | 88 | 87 | 88 | 82 | 75 | 91 | 86 | 103
  Week 52: Antihypertensive medication (Decreased) | 3 | 3 | 8 | 6 | 10 | 6 | 7 | 3 | 6
  Week 52: Antihypertensive medication (No change): number analyzed (Participants) | 77 | 88 | 87 | 88 | 82 | 75 | 91 | 86 | 103
  Week 52: Antihypertensive medication (No change) | 68 | 74 | 76 | 75 | 70 | 64 | 80 | 74 | 89
  Week 52: Antihypertensive medication (Increased): number analyzed (Participants) | 77 | 88 | 87 | 88 | 82 | 75 | 91 | 86 | 103
  Week 52: Antihypertensive medication (Increased) | 4 | 9 | 2 | 6 | 2 | 5 | 4 | 8 | 6
  Week 52: Antihypertensive medication (Missing): number analyzed (Participants) | 77 | 88 | 87 | 88 | 82 | 75 | 91 | 86 | 103
  Week 52: Antihypertensive medication (Missing) | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 2
  Week 0: Lipid-lowering medication (Yes) | 20 | 17 | 13 | 15 | 22 | 20 | 13 | 25 | 28
  Week 0: Lipid-lowering medication (No) | 83 | 85 | 90 | 88 | 80 | 82 | 90 | 78 | 108
  Week 52: Lipid-lowering medication (Decreased): number analyzed (Participants) | 77 | 88 | 87 | 88 | 82 | 75 | 91 | 86 | 103
  Week 52: Lipid-lowering medication (Decreased) | 0 | 1 | 3 | 1 | 1 | 3 | 3 | 1 | 2
  Week 52: Lipid-lowering medication (No change): number analyzed (Participants) | 77 | 88 | 87 | 88 | 82 | 75 | 91 | 86 | 103
  Week 52: Lipid-lowering medication (No change) | 73 | 83 | 81 | 84 | 79 | 71 | 87 | 83 | 94
  Week 52: Lipid-lowering medication (Increased): number analyzed (Participants) | 77 | 88 | 87 | 88 | 82 | 75 | 91 | 86 | 103
  Week 52: Lipid-lowering medication (Increased) | 2 | 2 | 2 | 2 | 2 | 1 | 1 | 1 | 5
  Week 52: Lipid-lowering medication (Missing): number analyzed (Participants) | 77 | 88 | 87 | 88 | 82 | 75 | 91 | 86 | 103
  Week 52: Lipid-lowering medication (Missing) | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 2

18. Secondary Outcome: Compliance With Nutritional Counselling
Description: This outcome measure presents "nutritional compliance results" recorded at weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52. Nutritional compliance was recorded on a 0 to 10 numeric rating scale (NRS), with higher scores representing better compliance.
Time Frame: Week 4-52
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 103 | 102 | 103 | 103 | 102 | 102 | 103 | 103 | 136
Score on a scale
  Week-4: number analyzed (Participants) | 97 | 99 | 100 | 98 | 99 | 96 | 101 | 101 | 131
  Week-4 | 6.85 (1.99) | 7.30 (1.96) | 7.17 (1.89) | 7.07 (2.27) | 7.20 (2.19) | 7.05 (2.02) | 7.30 (1.84) | 7.21 (2.13) | 6.08 (2.32)
  Week-8: number analyzed (Participants) | 97 | 98 | 95 | 96 | 96 | 89 | 99 | 97 | 124
  Week-8 | 6.53 (2.28) | 7.24 (1.91) | 6.82 (2.06) | 7.13 (2.03) | 7.00 (2.16) | 7.25 (1.84) | 7.65 (1.76) | 6.92 (2.18) | 5.85 (2.44)
  Week-12: number analyzed (Participants) | 94 | 93 | 91 | 95 | 95 | 83 | 94 | 95 | 118
  Week-12 | 6.70 (2.13) | 7.26 (2.26) | 7.22 (2.05) | 7.04 (2.17) | 7.11 (2.26) | 7.35 (1.96) | 7.64 (1.71) | 7.01 (1.93) | 6.14 (2.44)
  Week-16: number analyzed (Participants) | 85 | 93 | 88 | 94 | 88 | 82 | 95 | 94 | 115
  Week-16 | 6.85 (2.08) | 7.22 (1.96) | 7.36 (1.92) | 7.04 (2.05) | 7.61 (1.87) | 7.27 (2.11) | 7.71 (1.66) | 6.98 (1.87) | 6.31 (2.33)
  Week-20: number analyzed (Participants) | 86 | 89 | 92 | 92 | 88 | 82 | 90 | 88 | 111
  Week-20 | 6.92 (2.01) | 7.20 (1.98) | 6.87 (2.10) | 7.14 (1.88) | 7.64 (1.68) | 7.24 (2.16) | 7.74 (1.47) | 6.85 (2.20) | 6.24 (2.27)
  Week-24: number analyzed (Participants) | 86 | 93 | 89 | 90 | 87 | 82 | 89 | 89 | 110
  Week-24 | 6.49 (2.25) | 7.14 (2.05) | 7.07 (2.16) | 7.17 (1.86) | 7.63 (1.76) | 7.05 (1.96) | 7.55 (1.86) | 6.69 (2.12) | 6.06 (2.45)
  Week-28: number analyzed (Participants) | 83 | 91 | 88 | 91 | 84 | 80 | 91 | 87 | 107
  Week-28 | 6.94 (2.04) | 7.54 (1.78) | 7.10 (2.04) | 7.11 (1.73) | 7.46 (1.94) | 7.53 (1.57) | 7.47 (1.90) | 6.69 (2.04) | 6.34 (2.27)
  Week-32: number analyzed (Participants) | 78 | 91 | 90 | 88 | 85 | 78 | 91 | 86 | 104
  Week-32 | 6.83 (2.12) | 6.97 (2.23) | 7.12 (1.93) | 7.07 (2.07) | 7.72 (1.76) | 7.13 (2.23) | 7.29 (1.91) | 6.94 (2.01) | 5.86 (2.13)
  Week-36: number analyzed (Participants) | 77 | 89 | 87 | 88 | 83 | 76 | 88 | 86 | 101
  Week-36 | 6.87 (1.94) | 7.12 (2.02) | 7.03 (2.28) | 6.86 (1.98) | 7.20 (2.02) | 7.33 (1.84) | 7.34 (1.57) | 6.63 (2.16) | 6.10 (2.20)
  Week-40: number analyzed (Participants) | 78 | 88 | 86 | 88 | 84 | 77 | 88 | 86 | 104
  Week-40 | 6.86 (1.96) | 6.88 (2.40) | 7.07 (2.05) | 7.03 (1.97) | 7.40 (1.89) | 7.01 (1.81) | 7.26 (1.87) | 6.52 (2.07) | 5.90 (2.10)
  Week-44: number analyzed (Participants) | 72 | 87 | 84 | 84 | 80 | 78 | 88 | 80 | 102
  Week-44 | 6.83 (1.82) | 6.95 (2.10) | 6.96 (1.92) | 6.96 (2.01) | 7.30 (2.13) | 6.87 (1.98) | 7.30 (1.98) | 6.60 (1.85) | 5.99 (2.08)
  Week-48: number analyzed (Participants) | 74 | 87 | 85 | 84 | 81 | 75 | 87 | 82 | 98
  Week-48 | 6.82 (2.08) | 7.05 (1.91) | 6.88 (2.00) | 6.92 (2.16) | 7.12 (2.31) | 7.01 (2.03) | 7.23 (1.78) | 6.01 (2.49) | 6.16 (2.23)
  Week-52: number analyzed (Participants) | 74 | 88 | 84 | 87 | 81 | 75 | 89 | 85 | 100
  Week-52 | 7.23 (1.69) | 7.22 (1.98) | 7.05 (2.04) | 6.85 (2.47) | 7.36 (2.22) | 7.36 (1.85) | 7.31 (2.02) | 6.87 (2.07) | 6.09 (2.39)

19. Secondary Outcome: Number of AEs During the Trial
Description: Adverse events (AEs) were recorded from week 0 to week 59. Results are based on the in-trial observation period which was defined as the period from randomisation to last contact with trial site.
Time Frame: Week 0-59
Population: Overall number of participants analyzed = SAS which included all participants receiving at least one dose of the randomised treatment.
Measure: Number; unit: Events
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 103 | 102 | 103 | 103 | 102 | 102 | 103 | 103 | 136
Events | 547 | 730 | 738 | 587 | 775 | 737 | 681 | 612 | 650

20. Secondary Outcome: Number of Hypoglycaemic Episodes During the Trial
Description: Hypoglycaemic episodes were identified by either: 1) Subject reporting of symptoms of hypoglycaemia (low blood sugar) or 2) fasting plasma glucose (FPG) values ≤3.9 mmol/L (70 mg/dL) from blood sampling at site visits. Hypoglycaemic episodes were recorded from week 0 to week 59. Results are based on the in-trial observation period which was defined as the period from randomisation to last contact with trial site.
Time Frame: Week 0-59
Population: as for outcome 19
Measure: Number; unit: Episodes
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 103 | 102 | 103 | 103 | 102 | 102 | 103 | 103 | 136
Episodes | 1 | 6 | 4 | 8 | 10 | 20 | 16 | 4 | 18

21. Secondary Outcome: Number of New and Ongoing Nausea, Vomiting, Diarrhoea, and Constipation Events by Week
Description: Presented results are the number of nausea, vomiting, diarrhoea, and constipation events recorded from week 0 to week 59. Results are based on the in-trial observation period which was defined as the period from randomisation to last contact with trial site.
Time Frame: Week 0-59
Population: as for outcome 19
Measure: Number; unit: Events
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 103 | 102 | 103 | 103 | 102 | 102 | 103 | 103 | 136
Events
  Nausea | 41 | 80 | 74 | 69 | 94 | 106 | 97 | 89 | 30
  Vomiting | 10 | 29 | 41 | 18 | 35 | 32 | 47 | 17 | 6
  Diarrhoea | 29 | 37 | 61 | 54 | 63 | 54 | 49 | 46 | 23
  Constipation | 15 | 27 | 33 | 25 | 35 | 23 | 34 | 30 | 7

22. Secondary Outcome: Nausea: Individual Scores of Nausea Questionnaire and Severity by NRS Score
Description: This outcome measure presents results recorded at week 52. If a participant experienced an event of nausea within 24 hours prior to a site visit, a nausea questionnaire had to be completed. Participants experiencing such events were to answer 5 different categories in the questionnaire ('duration of nausea', 'time from the latest injection of trial product to the onset of nausea', 'time from last food intake to the onset of nausea', 'nausea accompanied by vomiting (yes/no)' and 'severity of nausea (worst during episode)'). Severity of nausea was recorded on a 0 to 10 numeric rating scale (NRS), where 0 = 'No nausea' and 10 = 'Nausea as bad as it could be'. Results are based on the in-trial observation period which was defined as the period from randomisation to last contact with trial site.
Time Frame: Week 52
Population: Overall number of participants analyzed = number of participants in the SAS who experienced an event of nausea within 24 hours prior to the site visit at week 52. SAS included all participants receiving at least one dose of the randomised treatment.
Measure: Number; unit: Events
Units Other Than Participants: Nausea events
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Number analyzed (Nausea events) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Events
  Duration of nausea:<30 min |  | 0 | 1 |  |  |  |  |  |
  Duration of nausea: 30 min-2 hr |  | 0 | 0 |  |  |  |  |  |
  Duration of nausea: 2-4 hr |  | 0 | 0 |  |  |  |  |  |
  Duration of nausea: 4-8 hr |  | 1 | 0 |  |  |  |  |  |
  Duration of nausea: >8 hr |  | 0 | 0 |  |  |  |  |  |
  Latest injection to onset time: 0-3 hr |  | 0 | 0 |  |  |  |  |  |
  Latest injection to onset time: 3-6 hr |  | 0 | 0 |  |  |  |  |  |
  Latest injection to onset time: 6-12 hr |  | 1 | 0 |  |  |  |  |  |
  Latest injection to onset time: 12-18 hr |  | 0 | 1 |  |  |  |  |  |
  Latest injection to onset time: >18 hr |  | 0 | 0 |  |  |  |  |  |
  Last food intake to onset time: 0-1 hr |  | 0 | 1 |  |  |  |  |  |
  Last food intake to onset time: 1-2 hr |  | 1 | 0 |  |  |  |  |  |
  Last food intake to onset time: 2-3 hr |  | 0 | 0 |  |  |  |  |  |
  Last food intake to onset time: 3-6 hr |  | 0 | 0 |  |  |  |  |  |
  Last food intake to onset time: >6 hr |  | 0 | 0 |  |  |  |  |  |
  Nausea accompanied by vomiting (Yes) |  | 0 | 0 |  |  |  |  |  |
  Nausea accompanied by vomiting (No) |  | 1 | 1 |  |  |  |  |  |
  Severity of nausea: 0 |  | 0 | 0 |  |  |  |  |  |
  Severity of nausea: 1 |  | 0 | 0 |  |  |  |  |  |
  Severity of nausea: 2 |  | 0 | 0 |  |  |  |  |  |
  Severity of nausea: 3 |  | 0 | 0 |  |  |  |  |  |
  Severity of nausea: 4 |  | 0 | 1 |  |  |  |  |  |
  Severity of nausea: 5 |  | 1 | 0 |  |  |  |  |  |
  Severity of nausea: 6 |  | 0 | 0 |  |  |  |  |  |
  Severity of nausea: 7 |  | 0 | 0 |  |  |  |  |  |
  Severity of nausea: 8 |  | 0 | 0 |  |  |  |  |  |
  Severity of nausea: 9 |  | 0 | 0 |  |  |  |  |  |
  Severity of nausea: 10 |  | 0 | 0 |  |  |  |  |  |

23. Secondary Outcome: Change in ECG
Description: Number of participants with electrocardiogram (ECG) results, "normal; abnormal, not clinically significant (NCS) or abnormal, clinically significant (CS)" was recorded at baseline (week 0) and week 52. Results are based on the on-treatment observation period which was defined as the period from first trial product administration to last trial product administration.
Time Frame: Week 0, week 52
Population: Overall number of participants analyzed = SAS which included all participants receiving at least one dose of the randomised treatment. Number Analyzed = number of participants in the SAS with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 103 | 102 | 103 | 103 | 102 | 102 | 103 | 103 | 136
Participants
  Week: 0: Normal | 70 | 69 | 74 | 62 | 62 | 70 | 74 | 68 | 85
  Week: 0: Abnormal, NCS | 33 | 31 | 29 | 41 | 38 | 32 | 27 | 35 | 51
  Week: 0: Abnormal, CS | 0 | 2 | 0 | 0 | 2 | 0 | 2 | 0 | 0
  Week: 52: number analyzed (Participants) | 82 | 91 | 87 | 89 | 87 | 77 | 92 | 86 | 106
  Week: 52: Normal | 57 | 73 | 67 | 58 | 57 | 55 | 64 | 59 | 66
  Week: 52: Abnormal, NCS | 25 | 18 | 18 | 31 | 29 | 21 | 28 | 26 | 40
  Week: 52: Abnormal, CS | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0

24. Secondary Outcome: Change in Pulse
Description: Change from baseline (week 0) in pulse rate was evaluated at week 52. Analysis of observed data using a mixed model for repeated measurements (MMRM) with treatment, region and sex as factors and baseline pulse as covariate, all nested within visit. Results are based on the on-treatment observation period which was defined as the period from first trial product administration to last trial product administration.
Time Frame: Week 0, week 52
Population: Overall number of participants analyzed = number of participants in the SAS with available data. SAS included all participants receiving at least one dose of the randomised treatment.
Measure: Least Squares Mean (Standard Error); unit: Beats per minute
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 101 | 102 | 103 | 103 | 102 | 102 | 103 | 103 | 135
Beats per minute | -0.33 (0.88) | 3.46 (0.83) | 1.88 (0.84) | 2.38 (0.83) | 2.54 (0.85) | 2.34 (0.89) | 2.15 (0.82) | 2.63 (0.84) | -0.86 (0.76)

25. Secondary Outcome: Change in Haematology: Haemoglobin
Description: Change from baseline (week 0) in haemoglobin was evaluated at week 52. Results are based on the on-treatment observation period which was defined as the period from first trial product administration to last trial product administration.
Time Frame: Week 0, week 52
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Millimoles per litre (mmol/L)
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 79 | 88 | 87 | 86 | 85 | 75 | 91 | 84 | 106
Millimoles per litre (mmol/L) | 0.01 (0.48) | -0.08 (0.65) | -0.02 (0.47) | -0.07 (0.51) | 0.00 (0.50) | -0.07 (0.47) | 0.02 (0.47) | 0.11 (0.48) | -0.01 (0.45)

26. Secondary Outcome: Change in Haematology: Haematocrit
Description: Change from baseline (week 0) in haematocrit was evaluated at week 52. Results are based on the on-treatment observation period which was defined as the period from first trial product administration to last trial product administration.
Time Frame: Week 0, week 52
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 79 | 88 | 87 | 86 | 85 | 75 | 91 | 84 | 106
Percentage of red blood cells | -0.25 (2.48) | -0.58 (3.28) | -0.42 (2.26) | -0.49 (2.67) | -0.31 (2.75) | -0.68 (2.82) | -0.15 (2.67) | 0.26 (2.70) | 0.26 (2.44)

27. Secondary Outcome: Change in Haematology: Thrombocytes, Leucocytes and Differential Count
Description: Change from baseline (week 0) in haematological parameters, "thrombocytes, leucocytes and differential cell count (eosinophils, neutrophils, basophils, monocytes and lymphocytes)" were evaluated at week 52. Results are based on the on-treatment observation period which was defined as the period from first trial product administration to last trial product administration.
Time Frame: Week 0, week 52
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: 10^9 cells/litre (L)
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 103 | 102 | 103 | 103 | 102 | 102 | 103 | 103 | 136
10^9 cells/litre (L)
  Thrombocytes: number analyzed (Participants) | 79 | 88 | 86 | 86 | 85 | 75 | 91 | 84 | 104
  Thrombocytes | -2.08 (35.26) | 2.95 (43.02) | -8.17 (42.59) | 2.79 (41.28) | -0.52 (39.59) | -5.76 (53.41) | -3.32 (45.02) | 4.83 (37.70) | -6.11 (39.11)
  Leucocytes: number analyzed (Participants) | 79 | 88 | 87 | 86 | 85 | 75 | 91 | 84 | 106
  Leucocytes | -0.47 (1.38) | -0.24 (1.44) | -0.23 (1.81) | -0.50 (1.42) | -0.68 (1.41) | -0.66 (1.90) | -0.40 (1.43) | -0.17 (1.41) | -0.44 (1.62)
  Eosinophils: number analyzed (Participants) | 79 | 88 | 87 | 86 | 85 | 73 | 91 | 84 | 106
  Eosinophils | 0.02 (0.11) | 0.02 (0.16) | -0.01 (0.09) | -0.02 (0.13) | 0.00 (0.08) | 0.01 (0.09) | -0.01 (0.08) | 0.01 (0.10) | 0.00 (0.08)
  Neutrophils: number analyzed (Participants) | 79 | 88 | 87 | 86 | 85 | 73 | 91 | 84 | 106
  Neutrophils | -0.36 (1.17) | -0.07 (1.22) | -0.05 (1.62) | -0.22 (1.24) | -0.51 (1.27) | -0.57 (1.76) | -0.23 (1.19) | -0.12 (1.11) | -0.33 (1.28)
  Basophils: number analyzed (Participants) | 79 | 88 | 87 | 86 | 85 | 73 | 91 | 84 | 106
  Basophils | 0.00 (0.03) | -0.00 (0.04) | -0.00 (0.03) | -0.01 (0.03) | -0.00 (0.03) | -0.01 (0.04) | 0.00 (0.04) | -0.00 (0.04) | 0.00 (0.04)
  Monocytes: number analyzed (Participants) | 79 | 88 | 87 | 86 | 85 | 73 | 91 | 84 | 106
  Monocytes | -0.04 (0.18) | -0.04 (0.12) | 0.01 (0.12) | -0.02 (0.10) | -0.02 (0.12) | -0.01 (0.13) | -0.03 (0.11) | -0.01 (0.14) | -0.02 (0.11)
  Lymphocytes: number analyzed (Participants) | 79 | 88 | 87 | 86 | 85 | 73 | 91 | 84 | 106
  Lymphocytes | -0.10 (0.36) | -0.16 (0.46) | -0.17 (0.38) | -0.24 (0.50) | -0.15 (0.36) | -0.08 (0.41) | -0.14 (0.37) | -0.06 (0.42) | -0.09 (0.66)

28. Secondary Outcome: Change in Haematology: Erythrocytes
Description: Change from baseline (week 0) in erythrocytes was evaluated at week 52. Results are based on the on-treatment observation period which was defined as the period from first trial product administration to last trial product administration.
Time Frame: Week 0, week 52
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: 10^12 cells/litre (L)
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 79 | 88 | 87 | 86 | 85 | 75 | 91 | 84 | 106
10^12 cells/litre (L) | -0.01 (0.26) | -0.06 (0.35) | -0.03 (0.27) | -0.04 (0.25) | -0.01 (0.29) | -0.04 (0.24) | -0.01 (0.27) | 0.05 (0.30) | 0.04 (0.24)

29. Secondary Outcome: Change in Biochemistry: Creatinine and Bilirubin (Total)
Description: Change from baseline (week 0) in biochemistry parameters, "creatinine and bilirubin (total)" were evaluated at week 52. Results are based on the on-treatment observation period which was defined as the period from first trial product administration to last trial product administration.
Time Frame: Week 0, week 52
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Micromole/litre (umol/L)
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 103 | 102 | 103 | 103 | 102 | 102 | 103 | 103 | 136
Micromole/litre (umol/L)
  Creatinine: number analyzed (Participants) | 79 | 88 | 87 | 88 | 85 | 76 | 92 | 86 | 105
  Creatinine | -1.14 (6.53) | -0.85 (7.59) | -1.09 (6.11) | 0.76 (8.11) | 1.48 (29.73) | 1.05 (8.45) | -2.10 (8.49) | -0.81 (7.16) | 0.28 (8.06)
  Bilirubin (total): number analyzed (Participants) | 79 | 88 | 87 | 87 | 85 | 76 | 92 | 85 | 105
  Bilirubin (total) | 0.30 (3.70) | 1.12 (3.60) | 1.59 (3.11) | 1.33 (3.61) | 1.23 (5.18) | 1.02 (4.04) | 1.67 (4.28) | 1.02 (3.67) | 1.09 (4.45)

30. Secondary Outcome: Change in Biochemistry: Creatinine Kinase, Amylase, Lipase, ALT, AST and ALP
Description: Change from baseline (week 0) in biochemistry parameters, "creatinine kinase, amylase, lipase, alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP)" were evaluated at week 52. Results are based on the on-treatment observation period which was defined as the period from first trial product administration to last trial product administration.
Time Frame: Week 0, week 52
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Unit/litre (U/L)
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 103 | 102 | 103 | 103 | 102 | 102 | 103 | 103 | 136
Unit/litre (U/L)
  Creatinine kinase: number analyzed (Participants) | 79 | 88 | 87 | 88 | 85 | 76 | 92 | 86 | 105
  Creatinine kinase | 0.53 (68.43) | -44.75 (266.88) | -13.20 (44.33) | -46.34 (163.09) | -29.91 (95.05) | -8.86 (47.28) | -28.08 (122.61) | -3.09 (172.46) | 53.36 (571.63)
  Amylase: number analyzed (Participants) | 79 | 88 | 87 | 88 | 85 | 76 | 92 | 86 | 105
  Amylase | 3.35 (13.82) | 4.84 (13.05) | 9.20 (12.72) | 7.53 (13.94) | 7.67 (16.26) | 8.39 (20.28) | 7.78 (14.82) | 7.12 (15.72) | 3.41 (12.27)
  Lipase: number analyzed (Participants) | 79 | 88 | 87 | 88 | 85 | 76 | 92 | 86 | 105
  Lipase | 5.62 (32.22) | 8.83 (28.10) | 17.55 (41.20) | 13.28 (34.86) | 13.33 (17.92) | 14.92 (44.31) | 15.09 (36.28) | 11.86 (27.48) | 1.63 (11.57)
  ALT: number analyzed (Participants) | 79 | 88 | 87 | 87 | 85 | 76 | 92 | 85 | 105
  ALT | -5.82 (20.97) | -5.45 (12.64) | -7.44 (17.14) | -9.15 (23.09) | -3.64 (11.30) | -9.07 (20.96) | -7.17 (12.62) | -2.95 (14.19) | -3.03 (11.91)
  AST: number analyzed (Participants) | 78 | 88 | 87 | 87 | 85 | 76 | 92 | 83 | 105
  AST | -1.08 (12.17) | -1.99 (7.95) | -2.33 (7.61) | -3.32 (10.22) | -2.07 (6.70) | -1.62 (10.78) | -2.73 (6.10) | -1.48 (10.13) | 0.00 (11.08)
  ALP: number analyzed (Participants) | 78 | 88 | 87 | 88 | 85 | 76 | 92 | 86 | 105
  ALP | -3.42 (13.04) | -3.44 (16.00) | -6.21 (10.96) | -6.70 (13.89) | -4.25 (12.65) | -3.50 (15.61) | -8.20 (14.13) | -0.52 (9.80) | -1.46 (11.39)

31. Secondary Outcome: Change in Biochemistry: Urea, Sodium, Potassium and Calcium (Total)
Description: Change from baseline (week 0) in biochemistry parameters, "urea, sodium, potassium and calcium (total)" were evaluated at week 52. Results are based on the on-treatment observation period which was defined as the period from first trial product administration to last trial product administration.
Time Frame: Week 0, week 52
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Millimole/litre (mmol/L)
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 103 | 102 | 103 | 103 | 102 | 102 | 103 | 103 | 136
Millimole/litre (mmol/L)
  Urea: number analyzed (Participants) | 79 | 88 | 87 | 88 | 85 | 76 | 92 | 86 | 105
  Urea | -0.04 (1.06) | 0.16 (1.26) | -0.01 (1.21) | -0.10 (1.25) | -0.00 (1.88) | -0.06 (1.33) | -0.33 (1.12) | 0.03 (1.06) | 0.21 (1.21)
  Sodium: number analyzed (Participants) | 79 | 88 | 87 | 88 | 85 | 76 | 92 | 86 | 105
  Sodium | -0.18 (2.47) | -0.27 (1.77) | -0.40 (2.41) | -0.82 (2.36) | -0.92 (2.62) | -0.76 (3.49) | -0.74 (2.71) | -0.37 (2.08) | -0.35 (2.08)
  Potassium: number analyzed (Participants) | 78 | 88 | 87 | 88 | 85 | 76 | 92 | 86 | 105
  Potassium | 0.01 (0.30) | 0.01 (0.38) | -0.00 (0.31) | -0.04 (0.36) | -0.10 (0.41) | 0.00 (0.36) | -0.11 (0.44) | -0.02 (0.35) | -0.04 (0.36)
  Calcium (total): number analyzed (Participants) | 79 | 88 | 87 | 88 | 85 | 76 | 92 | 86 | 105
  Calcium (total) | 0.01 (0.07) | -0.01 (0.09) | 0.01 (0.08) | 0.01 (0.08) | 0.00 (0.09) | -0.00 (0.08) | 0.00 (0.09) | 0.02 (0.08) | -0.00 (0.08)

32. Secondary Outcome: Change in Biochemistry: Albumin
Description: Change from baseline (week 0) in albumin was evaluated at week 52. Results are based on the on-treatment observation period which was defined as the period from first trial product administration to last trial product administration.
Time Frame: Week 0, week 52
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Gram/decilitre (g/dL)
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 79 | 88 | 87 | 88 | 85 | 76 | 92 | 86 | 105
Gram/decilitre (g/dL) | 0.03 (0.18) | 0.01 (0.21) | 0.07 (0.20) | 0.05 (0.21) | 0.03 (0.22) | 0.01 (0.21) | 0.02 (0.23) | 0.06 (0.18) | 0.04 (0.20)

33. Secondary Outcome: Change in Biochemistry: Calcitonin
Description: Change from baseline (week 0) in calcitonin was evaluated at week 52. Results are based on the on-treatment observation period which was defined as the period from first trial product administration to last trial product administration.
Time Frame: Week 0, week 52
Population: Overall number of participants analyzed = number of female participants in the SAS with available data. SAS included all participants receiving at least one dose of the randomised treatment.
Measure: Mean (Standard Deviation); unit: Nanogram/litre (ng/L)
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 54 | 55 | 54 | 56 | 58 | 47 | 59 | 57 | 64
Nanogram/litre (ng/L) | 0.08 (0.71) | 0.03 (1.07) | 0.04 (0.44) | 0.04 (0.18) | 0.17 (0.79) | -0.01 (0.73) | 0.20 (0.72) | 0.29 (1.27) | -0.12 (2.16)

34. Secondary Outcome: Change in Biochemistry: TSH
Description: Change from baseline (week 0) in thyroid stimulating hormone (TSH) was evaluated at week 52. Results are based on the on-treatment observation period which was defined as the period from first trial product administration to last trial product administration.
Time Frame: Week 0, week 52
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Milli-international units/litre (mIU/L)
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 79 | 88 | 86 | 88 | 85 | 76 | 92 | 86 | 105
Milli-international units/litre (mIU/L) | -0.31 (1.62) | -0.10 (1.10) | -0.22 (0.85) | -0.18 (1.04) | -0.10 (0.96) | -0.12 (0.84) | -0.43 (1.01) | 0.02 (0.88) | -0.07 (0.97)

35. Secondary Outcome: Change in Mental Health Assessed by C-SSRS
Description: Presented results are the number of participants with Columbia Suicidality Severity Rating Scale (C-SSRS) results recorded during baseline (week 0) and post baseline (week 4-52) visits. For classification of the events reported on the C-SSRS, the following categories were used: 1) Suicidal ideation, 2) Suicidal behaviour and 3) Non-suicidal self-injurious behaviour. Results are based on the on-treatment observation period which was defined as the period from first trial product administration to last trial product administration.
Time Frame: Week 0 and Week 4-59
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 103 | 102 | 103 | 103 | 102 | 102 | 103 | 103 | 136
Participants
  Wk 0: Suicidal ideation: number analyzed (Participants) | 102 | 102 | 103 | 103 | 102 | 102 | 103 | 103 | 136
  Wk 0: Suicidal ideation | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
  Wk 0: Suicidal behaviour: number analyzed (Participants) | 102 | 102 | 103 | 103 | 102 | 102 | 103 | 103 | 136
  Wk 0: Suicidal behaviour | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Wk 0: Non-suicidal self-injurious behaviour: number analyzed (Participants) | 102 | 102 | 103 | 103 | 102 | 102 | 103 | 103 | 136
  Wk 0: Non-suicidal self-injurious behaviour | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Wk 4-59: Suicidal ideation: number analyzed (Participants) | 100 | 102 | 102 | 102 | 102 | 102 | 103 | 103 | 134
  Wk 4-59: Suicidal ideation | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 1
  Wk 4-59: Suicidal behaviour: number analyzed (Participants) | 100 | 102 | 102 | 102 | 102 | 102 | 103 | 103 | 134
  Wk 4-59: Suicidal behaviour | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Wk 4-59: Non-suicidal self-injurious behaviour: number analyzed (Participants) | 100 | 102 | 102 | 102 | 102 | 102 | 103 | 103 | 134
  Wk 4-59: Non-suicidal self-injurious behaviour | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

36. Secondary Outcome: Change in Mental Health Assessed by PHQ-9
Description: Patient health questionnaire-9 (PHQ-9) was recorded at baseline (week 0) and week 52. The PHQ-9 questionnaire is a 9-item depression module included in the patient health questionnaire, a self-administered diagnostic tool used for assessment of mental disorders. On the PHQ-9, the participant rates the frequency of 9 items on a scale from 0 (not at all) to 3 (nearly every day). The PHQ-9 total score ranges from 0-27; total scores of 1-4 represent no depression, total scores of 5-9 represent mild depression, total scores of 10-14 represent moderate depression, total scores of 15-19 represent moderately severe depression and total scores of 20-27 represent severe depression. Results are based on the on-treatment observation period which was defined as the period from first trial product administration to last trial product administration.
Time Frame: Week 0, week 52
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
Number analyzed (Participants) | 103 | 102 | 103 | 103 | 102 | 102 | 103 | 103 | 136
Score on a scale
  Week 0 | 2.5 (3.4) | 1.7 (2.1) | 2.1 (2.6) | 1.5 (1.9) | 2.5 (2.9) | 1.7 (2.6) | 2.0 (2.2) | 2.0 (2.5) | 2.5 (3.1)
  Week 52: number analyzed (Participants) | 77 | 88 | 87 | 87 | 81 | 75 | 90 | 86 | 103
  Week 52 | 1.5 (2.2) | 1.1 (1.8) | 1.3 (2.0) | 1.1 (1.7) | 1.0 (1.8) | 1.1 (1.4) | 0.9 (1.6) | 1.3 (2.0) | 1.7 (2.6)

37. Secondary Outcome: Anti-semaglutide Antibodies During and After Treatment
Description: Participants were tested for anti-semaglutide antibodies from week 0 (post treatment) to week 52 (at weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52). This outcome measure is applicable only for the semaglutide treatment arms.
Time Frame: Week 0-52
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation)
Number analyzed (Participants) | 103 | 102 | 103 | 103 | 102 | 102 | 103
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Week 0 up to Week 59 (treatment period: week 0 to week 52 + follow-up period: week 53 to week 59).
Description: All AEs mentioned here are treatment-emergent adverse events (TEAEs), which was defined as any AE reported after first trial product administration and until last trial product administration with a 7-week follow-up period. Results are based on the safety analysis set, which included all subjects receiving at least 1 dose of randomised treatment.
Arm/Group | Semaglutide 0.05 mg | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.3 mg | Semaglutide 0.4 mg | Semaglutide 0.3 mg (Fast Escalation) | Semaglutide 0.4 mg (Fast Escalation) | Liraglutide 3.0 mg | Placebo Pool
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/102 | 0/103 | 0/103 | 0/102 | 0/102 | 1/103 | 0/103 | 0/136
Serious Adverse Events (participants affected / at risk) | 13/103 | 8/102 | 5/103 | 6/103 | 13/102 | 6/102 | 7/103 | 4/103 | 11/136
Other Adverse Events (participants affected / at risk) | 83/103 | 87/102 | 84/103 | 85/103 | 90/102 | 91/102 | 88/103 | 83/103 | 87/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 0.05 mg (N=103) | Semaglutide 0.1 mg (N=102) | Semaglutide 0.2 mg (N=103) | Semaglutide 0.3 mg (N=103) | Semaglutide 0.4 mg (N=102) | Semaglutide 0.3 mg (Fast Escalation) (N=102) | Semaglutide 0.4 mg (Fast Escalation) (N=103) | Liraglutide 3.0 mg (N=103) | Placebo Pool (N=136)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis Escherichia coli (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Human chorionic gonadotropin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infectious colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal scarring (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Percutaneous coronary intervention (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular insufficiency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Very long-chain acyl-coenzyme A dehydrogenase deficiency (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 0.05 mg (N=103) | Semaglutide 0.1 mg (N=102) | Semaglutide 0.2 mg (N=103) | Semaglutide 0.3 mg (N=103) | Semaglutide 0.4 mg (N=102) | Semaglutide 0.3 mg (Fast Escalation) (N=102) | Semaglutide 0.4 mg (Fast Escalation) (N=103) | Liraglutide 3.0 mg (N=103) | Placebo Pool (N=136)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 3 (3) | 6 (7) | 2 (2) | 3 (4) | 6 (6) | 4 (5) | 3 (3) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 7 (8) | 4 (6) | 2 (2) | 6 (7) | 8 (10) | 6 (7) | 6 (7) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (8) | 3 (6) | 16 (18) | 8 (10) | 9 (11) | 8 (8) | 5 (5) | 4 (5) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 4 (4) | 6 (6) | 6 (6) | 4 (5) | 6 (7) | 9 (14) | 5 (7) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 6 (6) | 1 (1) | 1 (1) | 6 (6) | 3 (3) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 6 (6) | 2 (3) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (9) | 9 (13) | 6 (7) | 4 (4) | 7 (8) | 4 (5) | 4 (6) | 5 (5) | 10 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (17) | 11 (16) | 6 (6) | 9 (10) | 3 (3) | 7 (7) | 8 (8) | 7 (7) | 10 (11)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 5 (7) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 4 (6) | 5 (5) | 4 (6) | 7 (7) | 3 (3) | 3 (3) | 2 (2) | 1 (2) | 9 (12)
Constipation (Gastrointestinal disorders) | 13 (15) | 22 (27) | 26 (33) | 18 (25) | 24 (35) | 19 (23) | 29 (34) | 24 (30) | 6 (7)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 2 (2) | 3 (3) | 4 (5) | 2 (2) | 1 (1) | 0 (0) | 7 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5) | 3 (3) | 6 (6) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 17 (17) | 13 (14) | 13 (14) | 14 (14) | 18 (21) | 20 (23) | 12 (13) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 20 (29) | 25 (37) | 35 (60) | 27 (54) | 38 (62) | 28 (52) | 28 (49) | 29 (46) | 16 (23)
Dizziness (Nervous system disorders) | 3 (3) | 6 (6) | 9 (9) | 4 (4) | 9 (11) | 8 (9) | 7 (8) | 7 (8) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 3 (5) | 8 (8) | 6 (8) | 14 (24) | 14 (17) | 15 (16) | 13 (19) | 8 (13) | 4 (5)
Early satiety (General disorders) | 3 (3) | 4 (4) | 5 (5) | 3 (3) | 6 (6) | 3 (3) | 3 (3) | 4 (4) | 2 (2)
Eructation (Gastrointestinal disorders) | 4 (4) | 8 (13) | 14 (20) | 8 (12) | 7 (7) | 17 (21) | 10 (12) | 6 (9) | 1 (1)
Fatigue (General disorders) | 4 (4) | 7 (7) | 7 (7) | 7 (7) | 13 (15) | 9 (10) | 7 (7) | 5 (6) | 9 (9)
Flatulence (Gastrointestinal disorders) | 4 (4) | 4 (4) | 3 (4) | 3 (3) | 6 (9) | 8 (10) | 5 (8) | 5 (6) | 3 (3)
Gastroenteritis (Infections and infestations) | 5 (7) | 11 (15) | 6 (6) | 8 (9) | 10 (11) | 4 (4) | 6 (6) | 4 (5) | 4 (6)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 (8) | 9 (9) | 8 (8) | 7 (8) | 10 (11) | 10 (13) | 9 (13) | 8 (9) | 0 (0)
Headache (Nervous system disorders) | 7 (9) | 15 (20) | 10 (12) | 10 (12) | 20 (31) | 14 (17) | 11 (13) | 15 (22) | 15 (19)
Influenza (Infections and infestations) | 2 (2) | 10 (14) | 4 (6) | 10 (13) | 2 (2) | 5 (5) | 7 (7) | 8 (9) | 8 (9)
Injection site bruising (General disorders) | 3 (4) | 5 (5) | 5 (8) | 5 (10) | 6 (6) | 5 (5) | 6 (8) | 4 (4) | 9 (27)
Insomnia (Psychiatric disorders) | 3 (3) | 6 (6) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Lipase increased (Investigations) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 6 (7) | 4 (4) | 1 (1) | 3 (4) | 1 (1)
Nasopharyngitis (Infections and infestations) | 16 (20) | 23 (26) | 19 (24) | 15 (20) | 19 (26) | 16 (18) | 20 (27) | 16 (22) | 16 (26)
Nausea (Gastrointestinal disorders) | 32 (41) | 42 (80) | 45 (74) | 43 (69) | 49 (94) | 55 (106) | 50 (97) | 46 (89) | 24 (30)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (9) | 3 (4) | 1 (1) | 4 (4) | 5 (6) | 4 (4) | 4 (5) | 7 (7)
Sinusitis (Infections and infestations) | 4 (6) | 5 (7) | 7 (10) | 3 (3) | 6 (6) | 5 (6) | 4 (6) | 6 (6) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 12 (16) | 10 (12) | 13 (17) | 10 (15) | 11 (16) | 10 (11) | 7 (8) | 12 (16) | 13 (19)
Urinary tract infection (Infections and infestations) | 3 (3) | 6 (6) | 4 (5) | 6 (6) | 2 (2) | 4 (5) | 3 (3) | 3 (3) | 5 (11)
Viral infection (Infections and infestations) | 5 (5) | 6 (8) | 3 (3) | 3 (3) | 4 (4) | 3 (3) | 4 (5) | 4 (4) | 4 (4)
Vomiting (Gastrointestinal disorders) | 8 (10) | 18 (29) | 24 (41) | 11 (18) | 17 (34) | 21 (32) | 23 (46) | 11 (17) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/11/NCT02453711/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/11/NCT02453711/SAP_001.pdf